CLINICAL TRIAL: NCT05343923
Title: Electrophysiological Substrate Characterization of Paroxysmal and Persistent Atrial Fibrillation: PAPER-AF Study
Brief Title: Atrial Fibrillation Characterization on Paroxysmal and Persistent Patients
Acronym: PAPER-AF
Status: Completed | Type: Observational
Sponsor: Felipe Atienza (Other)
Responsible Party: Sponsor-Investigator, Felipe Atienza, head of section (Cardiology Department), Hospital General Universitario Gregorio Marañon
Organization: Hospital General Universitario Gregorio Marañon (Other)
Other Study IDs: PI20/01618
Record Dates: First submitted 2021-05-19; First posted 2022-04-25 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- paroxistical AF
- persistent AF

SUMMARY:
Background and Hypothesis: Atrial Fibrillation (AF) treatment strategies have limitations. The efficacy of the procedure depends in several factors such as age, AF duration, atrial diameter and atrial electrophysiological behavior, determining what has been termed as atrial substrate. Therefore, the effectiveness of one specific treatment such as the ablation procedure, will be determined by the areas responsible for the maintenance of the fibrillation and its modification and/or elimination. The identification of these areas with a clear description of the arrhythmic substrate is one of the most important factors to determine new biomarkers that explain, at electrophysiological level, the properties of the substrate and therefore, increase the acute efficacy and long-term effectiveness of the treatment.

DETAILED DESCRIPTION:
The main objective of this project is to develop and validate new biomarkers based on a pre-existing methodology for the non-invasive identification of the mechanisms that are responsible for the maintenance of AF. This will be achieved by using a body surface potential mapping recording and using the signal to develop a new algorithm that is able to, from the acquired signals acquired during sinus rhythm, extract relevant features for an accurate prediction of long-term ablation outcome for patients with AF.

ELIGIBILITY:
Inclusion Criteria:

* Patients with paroxysmal or persistent AF symptomatic and refractory to at least one antiarrhythmic medication arriving in sinus rhythm to the electrophysiology laboratory.
* Patients must be able and willing to provide written informed consent to participate in the study.
* Prior anticoagulation for> 4 weeks or transesophageal echocardiogram excluding intracardiac thrombi.

Exclusion Criteria:

* Patients with inadequate anticoagulation levels, left atrial thrombus, tumor, or another abnormality which precludes catheter introduction on TEE prior to the procedure.
* Patients with moderate-to-severe mitral regurgitation.
* Patients with contraindications to systemic anticoagulation with heparin or coumadin.
* Patients who are or may potentially be pregnant.
* Current enrollment in another investigational drug or device study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with paroxysmal or persistent AF, arriving in sinus rhythm, undergoing catheter ablation (CA) procedure in the Gregorio Marañón Hospital between June 2021 and December 2023, will be included in this prospective study.
Sampling Method: Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Analysis of the signals on ECG during sinus rhythm | measurement will be performed at the inclusion point [0 months]
  measuring P-wave maximum value [milivolts]

SECONDARY OUTCOMES:
Analysis of the signals on ECG during sinus rhythm | 1) measurement will be performed at the inclusion point [0 months]
  measuring P-wave duration [miliseconds]

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital General Universitario Gregorio Marañón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided